CLINICAL TRIAL: NCT02692157
Title: NT-814: Evaluation of Its Ability to Alter the Abuse Liability of Oxycodone in an Exploratory Clinical Study
Acronym: NT-814
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was discontinued by the sponsor. No results to report
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Sandra D. Comer, Professor of Neurobiology, New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB#7173; U54DA037842 (NIH)
Record Dates: First submitted 2016-02-18; First posted 2016-02-25 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo Comparator: Placebo - During this arm, Placebo medication will be administered orally each evening at 8pm.
  Interventions: Drug: Placebo
- NT-814 50 mg (Active Comparator): Active Comparator: NT-814 50 mg - During this arm, 50 mg NT-814 will be administered orally each evening at 8pm.
  Interventions: Drug: NT-814 50 mg
- NT-814 100 mg (Active Comparator): Active Comparator: NT-814 100 mg - During this arm, 100 mg NT-814 will be administered orally each evening at 8pm.
  Interventions: Drug: NT-814 100 mg
- NT-814 200 mg (Active Comparator): Active Comparator: NT-814 200 mg - During this arm, 200 mg NT-814 will be administered orally each evening at 8pm.
  Interventions: Drug: NT-814 200 mg

INTERVENTIONS:
Drug: Placebo — Placebo for Neurokinin 1,3 antagonist
  Other Names: No other names
  Arms: Placebo
Drug: NT-814 50 mg — Neurokinin 1,3 antagonist 50 mg
  Other Names: GSK1144814 50 mg
  Arms: NT-814 50 mg
Drug: NT-814 100 mg — Neurokinin 1,3 antagonist 100 mg
  Other Names: GSK1144814 100 mg
  Arms: NT-814 100 mg
Drug: NT-814 200 mg — Neurokinin 1,3 antagonist 200 mg
  Other Names: GSK1144814 200 mg
  Arms: NT-814 200 mg

SUMMARY:
Healthy adult men who abuse opioids and are physically dependent on them will be invited to participate in a study to examine the ability of NT-814, a neurokinin (NK) antagonist at the 1 and 3 receptor subtypes, to alter the abuse liability of oxycodone.

DETAILED DESCRIPTION:
After completing the screening process, participants will be scheduled for admission onto the General Clinical Research Unit on 5-South for a 13-week study. During Week 1, participants will be detoxified from opioids. During Week 2 after the detoxification period, participants will be randomized to receive one of four maintenance doses of NT-814. During Weeks 3-4 participants may receive oxycodone during laboratory sessions and will complete a cue exposure session involving presentation of neutral and drug cues. Participants then will have the opportunity to self-administer drug by making clicks on a computer mouse. Weeks 2, 5, 8, and 11 will be medication stabilization weeks following by testing during Weeks 3-4, 6-7, 9-10, and 12-13. At the conclusion of the study, participants will be given an exit interview during which the study will be described. Those who are interested in treatment for their drug use at the end of the study will be offered referrals to studies at our Substance Treatment and Research Service or other treatment providers.

ELIGIBILITY:
Inclusion Criteria:

* DSM V criteria for Opioid Use Disorder moderate-severe (304.00)
* Physically healthy
* Able to perform study procedures
* Normal body weight (BMI <30 and >17.5), and total body weight >50 kg (110 lbs)
* Total testosterone in the laboratory normal range (250-1100 ng/dl)
* Current or history of intranasal opioid use.
* Must be willing to use adequate forms of contraception (e.g. condoms in combination with spermicide) for the duration of the study and a specified amount of time after participation.

Exclusion Criteria:

* On parole or probation
* Elevated liver function (i.e. AST and ALT >2 times the upper limit of normal) or impaired renal function (creatinine within normal limits)
* 12-lead ECG-based repeated demonstration of QTcF > 450 msec at screening
* HIV positive
* Any physical disorders that might make participation hazardous

Ages: 21 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Percentage of oxycodone choices | 1 week
  Percentage of drug (versus money) choices in each study arm will be our primary outcome measure.
Average visual analog scale ratings of "I like the choice" | 1 week
  Average ratings of oxycodone liking in each study arm will be obtained.

SECONDARY OUTCOMES:
Average visual analog scale ratings of "I want heroin" | 1 week
  Average ratings of "I want heroin" in each study arm will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra D Comer, PhD, Principal Investigator — NYSPI and Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via posters and talks at local and national conferences, as well as in publication form. The sharing of raw data will be done by request only, providing that there is a justifiable reason with a clear hypothesis and data analysis plan.

DOCUMENTS (2):
  • Study Protocol (2016-02-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT02692157/Prot_000.pdf
  • Statistical Analysis Plan (2016-02-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT02692157/SAP_001.pdf